CLINICAL TRIAL: NCT05953844
Title: Adherence to Antiretroviral Therapy in HIV Infected Individuals in Assiut Governorate, Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Sayed Sabra, doctor, Assiut University
Other Study IDs: HIV/AIDs
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Egypt is a HIV low prevalence country but between 2010 and 2019 newly infected cases have more than quadrupled, and the rise continues at an alarming pace. Maintaining over 95% adherence level among the PLHIV in developing countries is a crucial issue to maintain viral suppression, to minimize HIV related morbidity and mortality. The present study aims to identify the level of adherence and the factors influencing adherence to ART in Assiut Governorate. To the best of our knowledge, no previous studies on adherence to antiretroviral therapy and its associated factors in HIV infected individuals were done in Egypt.

DETAILED DESCRIPTION:
Egypt is a HIV low prevalence country but between 2010 and 2019 newly infected cases have more than quadrupled, and the rise continues at an alarming pace. According to the WHO country profile in 2021, 65% of people living with HIV (PLHIV) know their status, there is no statistic on viral load suppression, or the level of adherence to treatment among those who are under care.

To achieve optimal results from Antiretroviral therapy (at least 95%), high levels of patient adherence to ART is essential. Therefore, enhancing ART coverage is a principal strategy to end HIV/AIDS.

Medication adherence, which can be defined as the extent to which a patient's medicine-taking behavior corresponds with agreed instructions from a health care provider, is essential for realizing the potential benefits of most medication-based treatment. Many patients, especially those with chronic diseases, experience difficulties in adhering to a recommended treatment plan. Medication non-adherence, with average rates of those affected being between 30 and 50%, is a major challenge in the real-life treatment of these patients .

Despite several advances in ART for human immunodeficiency virus in the last decades, non-adherence continues to be a critical phenomenon in the treatment of these patients. Not only short-term virological response will be poor, but low drug concentrations also dramatically accelerate development of drug-resistance. So, maintaining over 95% adherence level among the PLHIV in developing countries is a crucial issue to maintain viral suppression, to minimize HIV related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* HIV +ve adults identified and listed by the HIV/AIDS National program in Assiut governorate.

Aged 18 years old and more.

Exclusion Criteria:

* prisoners children patients aged less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV +ve adults identified and listed by the HIV/AIDS National program in Assiut governorate.
Sampling Method: Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Extent of adherence to antiretroviral treatment | 6 MONTHS
  report on the extent of adherence to treatment by HIV +ve patients in Assiut Governorate.

SECONDARY OUTCOMES:
factors influencing adherence to ART | 6 months
  identification of factors influencing adherence to ART among HIV infected individuals in Assiut Governorate.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Result] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859
- [Result] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Result] Chesney MA. Factors affecting adherence to antiretroviral therapy. Clin Infect Dis. 2000 Jun;30 Suppl 2:S171-6. doi: 10.1086/313849. PMID 10860902
- [Result] Bangsberg DR, Perry S, Charlebois ED, Clark RA, Roberston M, Zolopa AR, Moss A. Non-adherence to highly active antiretroviral therapy predicts progression to AIDS. AIDS. 2001 Jun 15;15(9):1181-3. doi: 10.1097/00002030-200106150-00015. No abstract available. PMID 11416722
- [Result] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Result] Schaecher KL. The importance of treatment adherence in HIV. Am J Manag Care. 2013 Sep;19(12 Suppl):s231-7. PMID 24495293
- [Result] Burch LS, Smith CJ, Anderson J, Sherr L, Rodger AJ, O'Connell R, Geretti AM, Gilson R, Fisher M, Elford J, Jones M, Collins S, Azad Y, Phillips AN, Speakman A, Johnson MA, Lampe FC. Socioeconomic status and treatment outcomes for individuals with HIV on antiretroviral treatment in the UK: cross-sectional and longitudinal analyses. Lancet Public Health. 2016 Nov;1(1):e26-e36. doi: 10.1016/S2468-2667(16)30002-0. PMID 28299369
- [Result] Abdulrahman SA, Ganasegeran K, Rampal L, Martins OF. Conceptual Framework for Investigating and Influencing Adherence Behavior among HIV-Positive Populations: An Applied Social Cognition Model. AIDS Rev. 2019 Aug 6;21(3):157-159. doi: 10.24875/AIDSRev.19000028. PMID 31386650